CLINICAL TRIAL: NCT04844307
Title: Comparing COVID-19 Inpatient Outcomes When Treated With a Twice-a-day 15- Minute PT Program Versus a Once-a-day-30-minute PT Program
Brief Title: Comparing Inpatient COVID-19 Outcomes in 2 Different PT Dosing Groups
Acronym: CCPT
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Upon further review it has come to the PI's attention that the study may want no longer be very effective since most of our Covid patients are being discharged pretty quickly now that the treatments are so effective.
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021-12937
Record Dates: First submitted 2021-03-23; First posted 2021-04-14 (Actual); Last update posted 2022-02-21 (Actual); Status verified 2022-02

CONDITIONS: COVID-19; Cardiopulmonary Disease; Weakness, Muscle; Hypoxia; Debility Due to Disease
MeSH Terms: conditions — COVID-19; Pulmonary Heart Disease; Muscle Weakness; Hypoxia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard PT group (Active Comparator): The standard PT group (control) will be receiving the standard 30 minute PT sessions 5 days a week. There will be no variations from standard inpatient PT treatment except that subjects may receive more days of PT than patients who are not participating in study.
  Interventions: Other: Standard PT
- Divided session PT group (Experimental): The divided session PT group (experimental) will be receiving 15 minute sessions twice a day, five days a week. The total number of minutes of PT time per day/week will be identical to the standard PT group, but divided into shorter and more frequent sessions.
  Interventions: Other: Shorter duration higher frequency PT

INTERVENTIONS:
Other: Shorter duration higher frequency PT — The standard PT session (30 mins) will be divided into two 15 minute sessions spread out during the day. Therefore, the total number of minutes of PT will not vary from the standard.
  Arms: Divided session PT group
Other: Standard PT — The standard PT session is 30 minutes once daily. It routinely involves exercises designed to strengthen and increase mobility of the patient such as bed mobility, transfers, and ambulation. In this study group there will be no variation from this standard treatment.
  Arms: Standard PT group

SUMMARY:
The objective of this study is to compare the effects of twice-a-day 15-minute sessions of inpatient physical therapy (PT) to the standard daily 30 minute sessions. The patient outcomes that will be evaluated will be length of stay, change in functional status, and disposition (home/acute rehab vs. subacute/LTAC/death) in patients admitted with COVID-19.

DETAILED DESCRIPTION:
The 2019 pandemic struck New York City hospitals early and aggressively. In rehabilitating inpatients during the early part of the pandemic, we learned that many of them were too affected by the COVID-19 illness to be able to tolerate the typical 30-minute daily session of physical therapy. At that time, the physical therapy (PT) staff often accommodated patients by dividing the typical 30 minute daily session into two 15 minute sessions in an effort to increase patient tolerance and participation. However, it was discovered at that time that literature was scarce on whether these divided PT sessions were equal or superior to the typical sessions. Nor was there any substantial literature on whether shorter duration higher frequency sessions were better tolerated by the inpatient. The purpose of this prospective randomized non-blinded controlled study is to compare outcomes of COVID inpatients receiving one 30 minute daily session of PT to patients receiving two 15 minute daily sessions of PT.

In order to obtain high quality data on level of mobility during hospitalization, two separate scoring systems will be used: The AMPAC and JH-HLM scores. These two scoring systems have been selected for their wide acceptance in both the physiatry and physical therapy communities, and due to having confirmed inter-rater reliability and validity. These scores will be calculated by the physical therapist on initial evaluation, and then again on every session up until discharge. The physical therapy team at this community hospital have already received extensive education on the utilization of both of these scoring tools.

The rationale for this study is to determine whether shorter duration (15 minute) higher frequency sessions (2x a day) are better tolerated than the standard 30-minute session. We hypothesize that shorter duration higher frequency sessions are superior to standard inpatient PT sessions in terms of patient tolerance and change in mobility scores from admission to discharge. Supporting evidence is based on previous observation and from a recent survey given to 19 physical therapists actively working with COVID-19 inpatients at White plains Hospital: Healthier patients have a higher tolerance of the 30 minute sessions, and sicker patients have a poor tolerance of the 30 minute sessions.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-89.
* positive COVID19 status as confirmed by at least one positive nasopharyngeal/oropharyngeal swab or chest CT.
* PT referral placed and patient seen by PT within 72 hours of admission.

Exclusion Criteria:

* Patients who were deemed unable to actively participate in therapy due to poor cognitive status or being medically unstable.
* Patients who are unable to give consent.
* Patient who are bedbound at baseline.
* Patient who are not fluent in English or Spanish (a Spanish version of consent form will be made available)?

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-10 (Estimated); Primary Completion 2022-02 (Estimated); Study Completion 2022-02 (Estimated)

PRIMARY OUTCOMES:
Patient tolerance | Through completion of study, an average of 1 year
  Patient tolerance will be recorded in minutes at end of each PT session in each group.
Change in mobility scores from admission to discharge | Through completion of study, an average of 1 year
  Mobility scores including Activity Measure for Post Acute Care (AMPAC) and Johns Hopkins Highest Level of Mobility (JH-HLM) will be recorded at end of each PT session. The change in scores from admission to discharge will be determined and recorded once patient is discharged.

SECONDARY OUTCOMES:
Disposition | Through completion of study, an average of 1 year
  Disposition possibilities include home, home with services, acute rehab, subacute rehab or skilled nursing facility, LTACH, transfer to another acute care hospital, hospice/home with hospice, expired.
Hospital Length of Stay | Through completion of study, an average of 1 year
  Total length of stay in the hospital will be determined based on date of admission and date of discharge from acute care hospital.

CONTACTS AND LOCATIONS:
Overall Officials: Anupama Kurra, MD, Principal Investigator — Montefiore Medical Center

IPD SHARING:
Plan to Share IPD: No